CLINICAL TRIAL: NCT06676774
Title: Effect of Intranasal Oxytocin on Emotion Recognition and Acute Psycho-Social Stress-induced Cortisol Increase in Patients With Central Diabetes Insipidus (Arginine Vasopressin Deficiency) and Healthy Controls - the OxyMOTION-Study
Brief Title: Effect of Intranasal Oxytocin on Emotion Recognition and Acute Psycho-Social Stress-induced Cortisol Increase in Patients With Central Diabetes Insipidus and Healthy Controls
Acronym: OxyMOTION
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-01152; kt24christcrain7
Record Dates: First submitted 2024-11-01; First posted 2024-11-06 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Arginine Vasopressin Deficiency; Diabetes Insipidus
Keywords: intranasal oxytocin
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic; Diabetes Insipidus

STUDY DESIGN:
Intervention Model Description: Case-control trial with randomized, placebo-controlled, double-blind, cross-over design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part B oxytocin - Part A oxytocin - Part A Placebo - Part B Placebo (Experimental): Part A will investigate the recognition of facial emotions & body expressions in a cross-over design with a two-week wash-out period between both study visits. Part B will investigate the response of cortisol to acute psychosocial stress (TSST) with an eight-week wash-out period between both study visits. The order of group assignment is as follows: 1. Part B oxytocin, 2. Part A oxytocin, 3. Part A placebo, 4. Part B placebo
  Interventions: Drug: Oxytocin nasal spray; Other: Placebo
- Part B oxytocin - Part A Placebo - Part A oxytocin - Part B Placebo (Experimental): Part A will investigate the recognition of facial emotions & body expressions in a cross-over design with a two-week wash-out period between both study visits. Part B will investigate the response of cortisol to acute psychosocial stress (TSST) with an eight-week wash-out period between both study visits. The order of group assignment is as follows: 1. Part B oxytocin, 2. Part A placebo, 3. Part A oxytocin, 4. Part B placebo
  Interventions: Drug: Oxytocin nasal spray; Other: Placebo
- Part B Placebo - Part A Placebo - Part A oxytocin - Part B oxytocin (Experimental): Part A will investigate the recognition of facial emotions & body expressions in a cross-over design with a two-week wash-out period between both study visits. Part B will investigate the response of cortisol to acute psychosocial stress (TSST) with an eight-week wash-out period between both study visits. The order of group assignment is as follows: 1. Part B placebo, 2. Part A placebo, 3. Part A oxytocin, 4. Part B oxytocin
  Interventions: Drug: Oxytocin nasal spray; Other: Placebo
- Part B Placebo - Part A oxytocin - Part A Placebo - Part B oxytocin (Experimental): Part A will investigate the recognition of facial emotions & body expressions in a cross-over design with a two-week wash-out period between both study visits. Part B will investigate the response of cortisol to acute psychosocial stress (TSST) with an eight-week wash-out period between both study visits. The order of group assignment is as follows: 1. Part B placebo, 2. Part A oxytocin, 3. Part A placebo, 4. Part B oxytocin
  Interventions: Drug: Oxytocin nasal spray; Other: Placebo

INTERVENTIONS:
Drug: Oxytocin nasal spray — Participants will be instructed on correctly applying the intranasal study medication and will self-administer a single dose of 24 IU oxytocin under the supervision of unblinded study personnel.
Other: Placebo — Participants will be instructed on correctly applying the intranasal study medication and will self-administer a single dose of placebo (0.9% normal saline) under the supervision of unblinded study personnel.

SUMMARY:
This study aims to investigate the potential beneficial effects of intranasal oxytocin compared to placebo on emotion recognition and acute psychosocial stress in patients with arginine vasopressin deficiency compared to matched healthy controls.

DETAILED DESCRIPTION:
Arginine vasopressin (AVP) and oxytocin are both nine-amino acid neuropeptides produced in the hypothalamus and are released into circulation from axon terminals projecting to the posterior pituitary. Disruption of the hypothalamic-pituitary axis due to inflammation, tumours, or head trauma may cause AVP deficiency, formerly known as central diabetes insipidus, a condition characterised by polyuria and polydipsia. Once diagnosed with AVP deficiency, desmopressin (AVP receptor 2 analogue) is prescribed to overcome polyuria and polydipsia symptoms. However, despite adequate treatment with desmopressin, patients often report residual psychological symptoms such as heightened anxiety, impairment in identifying and expressing emotions, lower levels of empathy, and increased stress-related behaviour. Oxytocin regulates complex socio-emotional functioning, including attachment and pair bonding, fear extinction, emotion recognition, and empathy. In line with this, oxytocin acts as a stress-buffering hormone as it reduces cortisol in response to stress and has anxiolytic effects. In addition to its release from axonal terminals, there is dendritic release of oxytocin into the brain, including key regions engaged in social-emotional behaviour such as the amygdala, hippocampus, insula. Specifically, it has been supposed that the prosocial effect of oxytocin might be secondary to an anxiolytic effect that involves modulation of amygdala responsivity and by improving emotion recognition. Due to the anatomical proximity, disruption of the AVP system leading to AVP deficiency could also disturb the oxytocin system leading to an additional oxytocin deficiency. Therefore, the psychopathological findings in patients may be caused by an additional oxytocin deficiency. Established pituitary provocation tests, however, failed to show a consistent increase in oxytocin levels. Several studies documented marked acute increases in circulating oxytocin levels in response to 3,4-methylenedioxymethamphetamine (MDMA, known as 'ecstasy') in healthy individuals explaining the empathic feelings and prosocial and anxiolytic effects of MDMA. Based on these results, the study team recently investigated MDMA as a novel provocation test for oxytocin deficiency in patients with AVP deficiency. The study team thereby demonstrated an additional oxytocin deficiency in patients with AVP deficiency using this novel stimulation test with MDMA. Results from this study demonstrate no or only minimal increase in oxytocin after MDMA intake in AVP deficiency while an almost 8-fold increase from baseline values in healthy controls. Acute oxytocin-induced effects under MDMA, such as increased trust, closeness, and openness to others, identification of facial emotions, and fear extinction, were significantly lower in patients compared to healthy controls. Based on this, the additional oxytocin deficiency could explain the psychopathology in patients. Given these data and evidence, oxytocin treatment to improve emotion recognition, decrease anxiety, and buffer effusive stress-induced cortisol increase would have great clinical implications. To date, the central effects of intranasal oxytocin in patients with AVP deficiency have not been addressed, and whether oxytocin administration in these patients can improve the psychological symptoms and provide a novel treatment option needs to be answered. Therefore, this case-control trial with randomized, placebo-controlled, double-blind, cross-over design aims to investigate the effects of a single dose of intranasal oxytocin compared to intranasal placebo on emotion recognition, and acute anxiety and cortisol in response to acute psychosocial stress in patients with AVP deficiency compared to healthy controls.

ELIGIBILITY:
Inclusion criteria healthy controls

1. Adult healthy volunteers
2. Matched for age, sex, BMI, and oestrogen replacement/menopause/hormonal contraceptives to patients.
3. No medication, except hormonal contraception

Inclusion criteria

1. Adult patients with a confirmed diagnosis of AVP deficiency based on accepted criteria6
2. Stable hormone replacement therapy for at least three months with desmopressin and, in case of additional anterior pituitary deficiencies, with the respective substitution therapies.

Exclusion criteria

1. Participation in a trial with investigational drugs within 30 days
2. Active substance use disorder within the last six months
3. Consumption of alcoholic beverages >15 drinks/week
4. Current or previous psychotic disorder (e.g., schizophrenia spectrum disorder)
5. Pregnancy and breastfeeding within the last eight weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Effect of oxytocin compared to placebo in patients with AVP deficiency compared to healthy controls on recognition of facial emotions/body expression | up to 4 weeks
  Differences between the placebo and oxytocin session will be assessed for each participant in correct recognition of facial emotions & body expressions assessed with the EmBody (emotion from body expressions) /EmFace (emotion from facial expressions) task of 3 or more score points (score range: 20-80) The EmBody and EmFace subtasks comprise each of 42 stimuli showing body or facial expressions of angry, happy, or neutral affect (14 clips per emotion, half in front view and half in half-profile side view from the left). Stimuli last 1.5 seconds at 24 frames per second and are geometrically and optically standardized to prevent biases induced by ethnic cues (e.g., hair or skin tone) or clothing. Item order is pseudorandom to prevent sequence effects and was determined using the following constraints: the same emotion is shown no more than twice in a row; the same view per emotion is not shown consecutively (i.e., no angry-front, angry-front).
Effect of oxytocin compared to placebo in patients with AVP deficiency compared to healthy controls cortisol in response to acute stress | up to 10 weeks
  Differences between the placebo and oxytocin session will be assessed for each participant in cortisol levels in response to acute psychosocial stress induced upon the TSST (Trier Social Stress Test) by 15% or more in the area under the cortisol response curve.
  Salivary cortisol will be measured (as a measure of unbound cortisol concentrations in plasma) before and upon the TSST. Blood cortisol will also be measured The TSST consists of an unprepared speech and mental arithmetic performed in front of an audience.
  Previous studies indicated that this stress protocol reliably induces a significant HPA (Hypothalamic-pituitary-adrenal)-axis activation, with 2- to 3-fold increases in free cortisol and subjective responses indicative of moderate stress in healthy individuals.

SECONDARY OUTCOMES:
Emotion recognition | up to 4 weeks
  -Percentage of correct classifications per emotion in Facial Emotional Recognition Task (FERT). The FERT assesses the recognition of basic emotions.
  The task includes 10 neutral faces and 160 faces that express one of four basic emotions with pictures, morphed between 0% (i.e., neutral) and 100% in 10% steps. Stimuli are shown in random order for 500 ms, followed by the rating screen, where participants have to indicate the correct emotion.
Empathy | up to 4 weeks
  -Level of direct, indirect, and cognitive empathy for positive and negative emotions in the Multifaceted Empathy Task (MET). MET is a computer-assisted test, which consists of 40 photographs that show people in emotionally charged situations. To measure emotional empathy subjects are asked to rate how much they feel for an individual in each scene and how much they are aroused by each scene on a 1-9-point scale. The 3 aspects are each tested with 20 stimuli with positive valence and 20 with negative valence, resulting in a total of 120 trials.
Subjective emotional response to acute stress | up to 10 weeks
  Acute anxiety levels using the STAI-S (State-Trait Anxiety Inventory). This is a questionnaire to determine general anxiety levels. Based on responses to 40 items, with scores ranging from 1 ("almost never") to 4 ("almost always"), a total score is calculated. The STAI has two sub-scales, the State-Anxiety Scale (20 items) and the Trait-Anxiety Scale (20 items). The State-Anxiety Scale evaluates the current state of anxiety, asking how respondents feel "right now," using items that measure subjective feelings of apprehension, tension, nervousness, worry, and activation/arousal of the autonomic nervous system. The Trait-Anxiety Scale evaluates relatively stable aspects of "anxiety proneness," including general states of calmness, confidence, and security. The total scores range from 20 to 80, with higher scores indicating more pronounced anxiety.
Heart rate (bpm) | up to 10 weeks
  Heart rate as an indicator for subjective autonomic response to acute stress
blood pressure (mmHG) | up to 10 weeks
  Blood pressure as an idicator for subjective autonomic response to acute stress

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland